CLINICAL TRIAL: NCT03105648
Title: Diagnostic and Prognostic Significance of Computerized Cytologic Morphometry of the Thyroid Neoplasm
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201603064RIPB
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Computerized Cytomorphometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- thyroid cancer
  Interventions: Other: computerized cytomorphometry
- benign thyroid nodules
  Interventions: Other: computerized cytomorphometry

INTERVENTIONS:
Other: computerized cytomorphometry — use computer program to analyse the characteristics of thyroid cells obtained by fine needle aspiration cytology examination

SUMMARY:
The prevalence of thyroid nodule is worldwide high. About 40% of normal population has thyroid nodules and about 5% are malignancy. It is important to differentiate malignancy from benign nodules because the management is completely different. Nowadays, the gold standard is fine needle aspiration cytology (FNAC) examination. The overall sensitivity and specificity is fair (~90%), but still has its limitation that some results are indeterminate in about 15% of the nodules. These obstacles are especially troublesome for papillary and follicular thyroid cancer that leads to delayed diagnosis, incomplete resection, and repeated operation. Preoperative evaluation of the prognosis is extraordinary important for cancer management. However, current prognostic scoring systems is only applicable after surgery. Hence, we urgently need a better risk-stratification system for individual-tailored treatment, and genetic-based computerized morphometry study seems to be the most realistic and promising one. The goal of this study is to propose a reliable method for diagnosis and prognosis of papillary thyroid cancer and follicular thyroid cancer through analyzing cellular morphologic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* patients who previously had received thyroid fine needle aspiration cytology examination

Exclusion Criteria:

* patients who are younger than 20 years old

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who previously had received thyroid fine needle aspiration cytology examination
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
cytomorphometry of the cells | 2016/4/20-2026/4/20
  cytologic characteristics of the cells

CONTACTS AND LOCATIONS:
Overall Officials: Shyang-Rong Shih, Ph.D., Principal Investigator — National Taiwan University Hospita
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No